CLINICAL TRIAL: NCT01510496
Title: Transition From Acute to Chronic Pain After Inguinal Hernia, Hysterectomy and Thoracotomy : Analysis of Risk Factors and Association With Genetic Polymorphisms
Brief Title: Transition From Acute to Chronic Pain After Inguinal Hernia, Hysterectomy and Thoracotomy: Analysis of Risk Factors and Association With Genetic Polymorphisms
Status: Completed | Type: Observational
Sponsor: Fundacion IMIM (Other)
Responsible Party: Principal Investigator, Antonio Montes, MD, Fundacion IMIM
Other Study IDs: GENDOLCAT
Record Dates: First submitted 2011-12-23; First posted 2012-01-16 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Postoperative Pain
Keywords: Chronic pain; genetic polymorphisms; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Hysterectomy; Thoracotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample collection Five milliliters of venous blood will be extracted from each patient with chronic pain; control samples will come from a DNA bank. All patients must have given their written consent to testing and storage.
  - Plasma DNA will be extracted with a BioRobot EZ1 Workstation (Qiagen).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients who had inguinal herniorraphy.
  Interventions: Procedure: Inguinal herniorraphy.
- Patients who had hysterectomy.
  Interventions: Procedure: Hysterectomy.
- Patients who had thoracotomy.
  Interventions: Procedure: Thoracotomy .

INTERVENTIONS:
Procedure: Inguinal herniorraphy. — Inguinal herniorraphy (non laparoscopic).
  Groups: Patients who had inguinal herniorraphy.
Procedure: Hysterectomy. — Hysterectomy: Vaginal and abdominal.
  Groups: Patients who had hysterectomy.
Procedure: Thoracotomy . — Thoracotomy (non laparoscopic).
  Groups: Patients who had thoracotomy.

SUMMARY:
The treatment of postoperative pain continues to be inadequate in the investigators practice setting.

Inadequate pain treatment not only contributes to postoperative complications in the short term but can also be a factor that favors the development of chronic postoperative pain and diminishes long-term quality of life. Risk factors that can lead to a transition to chronic pain need to be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with given inform consent, aged mor than 18 years, who undergo scheduled surgery of one of the following types: inguinal hernia (men), hysterectomy, thoracotomy (men).

Exclusion Criteria:

* Patients aged less than 18 years,
* Patients requiring reoperation because of surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All spanish patients who undergo scheduled surgery of one of the following types: inguinal herniorrhaphy, hysterectomy, toracothomy.
Sampling Method: Non-Probability Sample
Enrollment: 3979 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of chronic postsurgical pain. | After 3 and 12 months of surgery.
  After 3 months a physical examination will take place and after 12 months a follow-up will be reported by phone.

SECONDARY OUTCOMES:
Predictive factors of chronic postsurgical pain. | After 3 and 12 months of surgery.
  Preoperative (psychological factors, preoperative pain, pharmacologic treatment) intraoperative (surgical technic, type of anaestesia) and postoperative(posoperative pain, surgical complications and treatment of postoperative pain).

CONTACTS AND LOCATIONS:
Locations (26):
- Spain (26):
  - Hospital Municipal de Badalona, Badalona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de l'Esperança, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Sagrat Cor, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital del Sant Boi, Barcelona, Barcelona
  - Hospital de San Bernabé, Berga, Barcelona
  - Hospital de Granollers, Granollers, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Manresa, Manresa, Barcelona
  - Hospital de Mataro, Mataró, Barcelona
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitari Mutua de Terrassa, Terrassa, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Universitari Doctor Josep Trueta de Girona, Girona, Girona
  - Hospital de Santa Caterina, Salt, Girona
  - Hospital Santa Maria, Lleida, Lleida
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari de la Fe, Valencia, Valencia
  - Hospital Lluís Alcanyís de Xàtiva, Xàtiva, València

REFERENCES:
- [Derived] Bande D, Molto L, Pereira JA, Montes A. Chronic pain after groin hernia repair: pain characteristics and impact on quality of life. BMC Surg. 2020 Jul 6;20(1):147. doi: 10.1186/s12893-020-00805-9. PMID 32631293
- [Derived] Montes A, Roca G, Sabate S, Lao JI, Navarro A, Cantillo J, Canet J; GENDOLCAT Study Group. Genetic and Clinical Factors Associated with Chronic Postsurgical Pain after Hernia Repair, Hysterectomy, and Thoracotomy: A Two-year Multicenter Cohort Study. Anesthesiology. 2015 May;122(5):1123-41. doi: 10.1097/ALN.0000000000000611. PMID 25985024